CLINICAL TRIAL: NCT00006037
Title: Phase II Randomized Placebo-Controlled Double-Blinded Study With 5-FU vs. 5-FU With IM862 With Cross-Over to CPT-11 vs. CPT-11 With IM862
Brief Title: Chemotherapy Plus IM-862 in Treating Patients With Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug not available
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000068052 (3C-99-3); LAC-USC-3C993; NCI-G00-1812
Record Dates: First submitted 2000-07-05; First posted 2004-02-26 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: oglufanide disodium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. IM-862 may stop the growth of colorectal cancer by stopping blood flow to the tumor. It is not yet known if chemotherapy is more effective with or without IM-862 in treating colorectal cancer.

PURPOSE: Randomized phase II trial to study the effectiveness of chemotherapy plus IM-862 in treating patients who have metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy of fluorouracil with or without IM-862 in terms of progression free survival in patients with previously untreated or recurrent metastatic adenocarcinoma of the colon or rectum. II. Determine the toxicity of IM-862 and fluorouracil in these patients. III. Determine the efficacy of IM-862 in combination with irinotecan in terms of progression free survival in patients who have disease progression after receiving fluorouracil. IV. Obtain preliminary data on molecular markers of response and time to progression by determining levels of genes involved in adhesion, angiogenesis, apoptosis, and drug resistance prior to and during chemotherapy. V. Determine the molecular correlates for response and time to progression through analysis of serum and urine markers of angiogenesis, such as vascular endothelial growth factor and fibroblast growth factor, in patients treated with IM-862 in combination with fluorouracil or irinotecan. VI. Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, double blind, placebo controlled, crossover study. Patients are randomized to one of two treatment arms: Arm I: Patients receive fluorouracil IV continuously on days 1-21 and IM-862 intranasally three times daily on days 1-28. Courses repeat every 4 weeks in the absence of disease progression. Patients who develop disease progression are taken off fluorouracil and IM-862, and then receive irinotecan IV over 90 minutes weekly for 4 weeks. Courses repeat every 6 weeks in the absence of disease progression. Arm II: Patients receive fluorouracil as in arm I and placebo intranasally three times daily on days 1-28. Courses repeat every 4 weeks in the absence of disease progression. Patients who develop disease progression are taken off fluorouracil and placebo, and then receive irinotecan and IM-862 as in arm I on days 1-42. Courses repeat every 6 weeks in the absence of disease progression. Quality of life is assessed prior to study, and then prior to every course during study. Patients are followed for a minimum of 6 months.

PROJECTED ACCRUAL: A total of 66 patients (33 per arm) will be accrued for this study within 26-27 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven metastatic adenocarcinoma of the colon or rectum Previously untreated OR Recurrent with a disease free period of at least 1 year Measurable or evaluable disease Tumor must be accessible for biopsy No brain metastasis

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: SWOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute granulocyte count greater than 1,000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin no greater than 2 times upper limit of normal (ULN) (no greater than 3 times ULN if liver metastasis present) AST or ALT no greater than 2 times ULN (no greater than 5 times ULN if liver metastasis present) Renal: Creatinine no greater than 1.25 times ULN Cardiovascular: No myocardial infarction within the past year No congestive heart failure Other: No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for at least 6 months after study No medical, social, or psychological factor that would interfere with compliance

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior adjuvant immunotherapy with monoclonal antibody 17-1A allowed No prior IM-862 Chemotherapy: At least 1 year since prior chemotherapy for patients with recurrent metastatic adenocarcinoma of the colon or rectum Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy No concurrent radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 1999-11; Primary Completion 2001-11 (Actual); Study Completion 2001-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heinz-Josef Lenz, MD, Study Chair — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California, United States